CLINICAL TRIAL: NCT02510768
Title: A Randomized, Within-Subject, Placebo-Controlled, Single-Blind Study to Evaluate the Efficacy of ELAPR002f and ELAPR002g in Women With Striae Distensae (SD) Alba
Brief Title: A Study to Evaluate the Efficacy of ELAPR in Women With Striae Distensae Alba
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elastagen Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ELAPR-P1C
Record Dates: First submitted 2015-07-26; First posted 2015-07-29 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Striae Distensae
Keywords: alba
MeSH Terms: conditions — Striae Distensae

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ELAPR002f (Experimental): ELAPR002f A tropoelastin polymer cross-linked with hyaluronic acid.
  Interventions: Device: ELAPR002f
- ELAPR002g (Experimental): ELAPR002g A tropoelastin polymer cross-linked with hyaluronic acid.
  Interventions: Device: ELAPR002g
- Saline (Placebo Comparator): Saline
  Interventions: Device: Saline

INTERVENTIONS:
Device: ELAPR002f — Intradermal implant
  Arms: ELAPR002f
Device: ELAPR002g — Intradermal implant
  Arms: ELAPR002g
Device: Saline — Intradermal implant
  Arms: Saline

SUMMARY:
The study is designed to evaluate the efficacy of two formulations of a cross-linked tropoelastin matrix given the product codes ELAPR002f and ELAPR002g (collectively referred to as ELAPR or ELAPR002) for the treatment of Striae Distensae (SD) alba when administered as intradermal implants.

DETAILED DESCRIPTION:
The study will consist of six study visits. There will be a screening visit to confirm eligibility and to assess baseline parameters (Day -28 to Day -1). For enrolled subjects there will be three intradermal (i.d.) treatment sessions of ELAPR002f or ELAPR002g and placebo, given at one-monthly intervals (approximately Day 0, Day 28 and Day 56). There will be a safety assessment visit 7 days after the first treatment session (Day 7) to review any adverse events and assess the implant sites. ELAPR002f or ELAPR002g will be administered alone vs. placebo. Subjects will be followed for a total of 12 weeks (to Day 84) following the first treatment, with efficacy and safety assessments undertaken at each study visit. At the final follow-up visit (Day 84) a biopsy sample will be taken from each of the treated SDs (active and placebo treated), together with a control biopsy of normal skin collected from an area of the lateral aspect of the abdomen, hip or thigh without an SD alba. Each study subject will act as their own control with active and placebo treatments given single-blind to contralateral sides of the abdomen, hip or thigh, into matched and paired SD. Prior to administration the selected injection sites along the length of SD alba to be treated will be identified and marked with a semi-permanent mark to ensure consistency of anatomic sites for treatment and biopsy. Follow-up period extended to D168, D336 and D504.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects with at least four abdominal, hip or thigh SD alba which are approximately bilaterally symmetrical (similar dimensions/location/colour) and are of at least 6 cm in length and no more than 5mm wide.
* SD alba within an area of skin of otherwise normal, smooth, mainly flat appearance.
* Age: 30 - 55 years.
* BMI: 18.5 to 35.0 Kg/m2.
* Capable of providing voluntary informed consent.
* Good general health.
* Female subjects who are sexually active will be of non-child bearing potential (i.e., surgically sterilized or postmenopausal), abstain from sexual intercourse, or use a reliable method of contraception (e.g. hormonal contraceptive, condom, IUD) for at least 30 days prior to dosing and during the duration of the study.
* Fitzpatrick skin types II, III or IV.

Exclusion Criteria:

* SD alba within an area of otherwise abnormal skin appearance including unusual lumpiness or abnormal skin laxity.
* Current or previous medical or surgical treatment of SD.
* Known hypersensitivity to tropoelastin, hyaluronic acid or any other component of ELAPR002f or ELAPR002g.
* Female subjects with a positive pregnancy test, women refusing to agree to adequate contraception and pregnancy tests during the study, or women who are planning to become pregnant during the period of the trial.
* Participation in a clinical trial of a pharmacological agent within 1 month prior to screening.
* Clinically significant haematology or biochemistry findings at screening.
* Positive test for hepatitis B, hepatitis C or HIV at screening.
* Bleeding diathesis, anticoagulant drugs, thrombocytopenia or clinically significant prolonged activated partial thromboplastin time (APTT) or prothrombin time (PT).
* Chronic use of aspirin, other non-steroidal anti-inflammatory drugs or other anti-platelet agents.
* History of keloid formation.
* Systemic corticosteroids within last 12 weeks.
* Diabetes or other metabolic disorders that may interfere with the subject's response to treatment in the opinion of the investigator.
* Any serious medical condition which in the opinion of the investigator would have a strong possibility of requiring systemic corticosteroid medication.
* Females who are pregnant or lactating.
* Previous administration of tropoelastin.
* A history of anaphylaxis or allergic reactions including any known hypersensitivity to lidocaine.
* Use of any investigational product on the intended implant site in the previous 12 months.
* Fitzpatrick skin types I, V or VI.
* Any other factor that in the opinion of the Investigator would make the subject unsafe or unsuitable for the study.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-04-16 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2018-03-06 (Actual)

PRIMARY OUTCOMES:
Size of SD alba scars pre and post treatment. | 3 months
  Measurement of scar dimensions pre and post treatment (width x length x depth in mm) as measured by 3D photography, also 2D photography, subject satisfaction and biopsy (histology).

SECONDARY OUTCOMES:
Frequency and severity of implant site reactions post treatment. | 3 months
  Measure incidence and severity of implant site reactions as assessed by clinical observation and subject diary card records.

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided